CLINICAL TRIAL: NCT01050335
Title: Collaborative Surgical Proficiency Initiative
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Phoenix Integrated Surgical Residency (Other)
Responsible Party: Kanav Kahol, PhD Principal Investigator, Simulation and Education Training (SimET) Center, Banner Good Samaritan Medical Center
Other Study IDs: 01-07-0044
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2009-06

CONDITIONS: Surgical Proficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical resident or attending
  Interventions: Behavioral: Simuvision Simulator

INTERVENTIONS:
Behavioral: Simuvision Simulator — Participants will perform common surgical procedures on the simulator

SUMMARY:
The purpose of this study is to provide a quantitative base line comparison to determine a surgeon's proficiency based on that surgeon's hand and tool movements while performing simulation tasks.

ELIGIBILITY:
Inclusion Criteria:

* Surgical residents and attendings from Banner Good Samaritan Medical Center
* Range in age from 23-65 years
* Willing to provide informed consent

Exclusion Criteria:

* N/A

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical residents and attendings from Banner Good Samaritan Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kanav Kahol, PhD, Principal Investigator — Simulation and Education Training (SimET) Center, Banner Good Samaritan Medical Center; John Ferrara, MD, Study Director — Phoenix Integrated Surgical Residency
Locations (1):
- Simulation and Education Training (SimET) Center, Banner Good Samaritan Medical Center, Phoenix, Arizona, United States